CLINICAL TRIAL: NCT01872000
Title: A Prospective Randomised Controlled Trial to Assess Improved Binocular Visual Function in Young Patients Undergoing Monocular Cataract Surgery With a Bifocal Intraocular Lens.
Brief Title: Binocular Vision in Monocular Pseudophakia
Acronym: BVMP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment.
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BVMP2013
Record Dates: First submitted 2013-05-01; First posted 2013-06-07 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2018-10

CONDITIONS: Cataract
Keywords: Intraocular lens; Phacoemulsification
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal IOL (Experimental): Phacoemulsification and IOL inserted following cataract surgery
  Interventions: Procedure: Cataract surgery
- Standard IOL (Active Comparator): Phacoemulsification and IOL inserted following cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery
  Other Names: Phacoemulsification and IOL insertion

SUMMARY:
Following cataract surgery, an intraocular lens (IOL) is implanted in the eye. The majority of people develop an operable cataract when they are over the age of 50. Occasionally people under 50 years develop a cataract requiring an operation. The visual demands in this age group are very different due to both physiological and lifestyle factors. Traditionally IOLs are focussed for distance vision and additional spectacles are worn for near vision. Under the age of 45 years we have the ability to naturally change the focus of our eyes and do not require additional reading glasses. This is known as accommodation. By removing the cataractous lens and replacing it with an IOL with a fixed single focus, both eyes work together for distance vision but only the unoperated eye is able to change focus for different working distances. This study aims to establish whether a multifocal IOL implanted in one eye is able to complement the accommodation in the other eye so the 2 eyes work more effectively together. This may enhance depth perception and improve the quality of vision. Depth perception is important for more comfortable vision on the computer screen, when reading and for jobs that require good depth perception.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 - 45.
* Cataract operation required in one eye only, either due to the presence of cataract affecting visual function, or in combination with surgery which is likely to cause visually significant cataract.
* Expected visual improvement in operable eye of at least 6/12.
* Fellow eye with a VA of at least 6/9.
* Astigmatism of 1.0D or less.
* Target of emmetropia in the operated eye.
* Intact posterior capsule with planned implantation into the capsular bag.
* IOL power required 10 - 30D.

Exclusion Criteria:

* Pre-existing amblyopia or squint.
* Significant diabetic retinopathy.
* Macular off retinal detachment with metamorphopsia or poor visual prognosis.
* Other macula or ophthalmic pathology affecting macula function resulting in poor visual prognosis.
* Pregnancy, lactating or planned pregnancy during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Extent of binocular vision at near working distance following IOL implantation. | 3-6 months

SECONDARY OUTCOMES:
Change in visual acuity and subjective visual comfort at distance, intermediate and near working distances following IOL implantation. | 3-6 months
  Visual acuity at different distances will be presented in combination as they are linked.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, DPhil, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Stoke Mandeville Hospital, Aylesbury